CLINICAL TRIAL: NCT04742868
Title: Recovery of Soccer Players After Anterior Cruciate Ligament Reconstruction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Carolina Fernández Lao, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGranada111
Record Dates: First submitted 2020-11-05; First posted 2021-02-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Knee Injuries and Disorders
Keywords: ACLR; Quadricepses tendon graft; hamstring tendon graft
MeSH Terms: conditions — Knee Injuries; Disease | interventions — Anterior Cruciate Ligament Reconstruction; Bone Transplantation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: the researcher will evaluate each patient without knowing the type of grafting that will be applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 QUADRICEPS TENDON WITH BONE GRAFT (Experimental): Quadriceps tendon with bone will be used as graft for the surgery.
  Interventions: Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH QUADRICEPS TENDON WITH BONE GRAFT; Other: Rehabilitation protocol
- Arm 2 HAMSTRING TENDON GRAFT (Experimental): Hamstring tendon with bone will be used as graft for the surgery
  Interventions: Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH HAMSTRING TENDON GRAFT; Other: Rehabilitation protocol
- Arm 3. QUADRICEPS TENDON WITHOUT BONE GRAFT (Experimental): Quadriceps tendon without bone will be used as graft for the surgery.
  Interventions: Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH QUADRICEPS TENDON WITHOUT BONE GRAFT; Other: Rehabilitation protocol

INTERVENTIONS:
Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH QUADRICEPS TENDON WITH BONE GRAFT — Quadriceps tendon with pattlar bone will used for grating
  Arms: Arm 1 QUADRICEPS TENDON WITH BONE GRAFT
Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH HAMSTRING TENDON GRAFT — Hamstring tendon with will used for grating
  Arms: Arm 2 HAMSTRING TENDON GRAFT
Procedure: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION WITH QUADRICEPS TENDON WITHOUT BONE GRAFT — Quadriceps tendon without pattlar bone will used for grating
  Arms: Arm 3. QUADRICEPS TENDON WITHOUT BONE GRAFT
Other: Rehabilitation protocol — All patients will receive six months rehabilitation program which aim to recover the strength and function

SUMMARY:
The purpose of this CRT study is to compare clinical and functional outcomes of three graft types ( Quadriceps tendon with bone versus Hamstring tendon versus Quadriceps tendon without bone) for reconstration of anterior cruciate ligament among football players.

DETAILED DESCRIPTION:
In the previous studies patellar tendon and hamstring tendon were the most investigated graft types. While quadriceps tendon has been investigated a fewer times. And to our knowledge there is no control study that compare quadriceps tendon-patellar bone autograft with Quadriceps Autograft and Hamstring Autograft as control randomized study.

All of the patients will be examined before of the surgery and 3, 6, 12, 24 months after the surgery to compare the outcome of differnt graft types. While a secand aim of this study is to examen the effect of rehabilitation protocol on the short and long term within all of the clinical and the functional outcomes.

The rehabilitation protocol will contain one phase before the surgery and four phases after the surgery.The goal of the first phase will be pain and inflammation control, increase ROM and muscle strength will be during the second and the third phases.In the last phase all of the players have to achieve maximum muscle strength and neuromuscular control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACL injury susceptible to receive a surgical reconstruction.
* Autograft with Hamstring tendon ,quadriceps tendon or quadriceps tendon with patellar bone.
* Soccer player for more than 3 years.
* Between 16 and 40 years old.

Exclusion Criteria:

* Patient with previous joint injury.
* Patient with previous surgery on the affected knee.
* patient with previous musculoskeletal injury (4 weeks)
* Patient with untreated chronic injury.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change of Isokinetic strenght test | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  the assessment will be made with GENU 3 dynamometer (GENU 3, Easytech, Firenze, Italy), using isokinetic parameters at angular velocities of 60°/sec (3 repetitions), 180°/sec (5 repetitions) and 300°/sec (15 repetitions) with 30 seconds of rest among these. To determine the height of the chair, the lateral femoral condyle was aligned with the rotational axis of the dynamometer. The peak torque, average torque and flexor-extensor torque rate value. Patients will be warm up in a cycle ergometer previously (5 min) and them performing mobilization exercises and stretching in lower limbs (5 min).

SECONDARY OUTCOMES:
Visual Analogical Scale | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  the participants will be completed a visual analogue scale (0-10 points) to assess the presence of knee pain.
Pressure Pain Thresholds | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  We will use an electronic algometer (Somedic AB, Farsta, Sweden) over 6 points: epicondyle (1), at the midpoint between the greater trochanter and the lateral condyle of the femur on the external (2), at three centimeters above the patella in the vastus medialis (3), at the midpoint between the lower pole of the patella and the anterior tuberosity of the tibia (4), at 3 cm above the patella in midline of the thigh (5) and at the inclusion of the goose leg. The mean of 3 trials will be used for the main analysis.
MUSCLE ARQUITECTURE | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  an ultrasound device (MyLab™ 25, Esaote Medical Systems,Genova, Italy) and a 12 MHz linear probe will be used in this study. The depth and width of quad tendon and articular cartilage of femoral trochlea will be captured.
ANTEROPOSTERIOR LAXITY | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  it will be measured using the KT-2000 TM arthrometer (MEDmetric, Sn Diego, CA, USA)
Tegner questionnaire | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  It is a subjective satisfaction index of on a scale of 0 to 100
Single-legged hop test | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  The patient is placed standing on one leg and must jump as far as possible landing on the same leg.

OTHER OUTCOMES:
Body Mass Index ) | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  in kg/m2, will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea
Fat mass | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  %fat mass will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)
Lean Mass | Patients will be examined before , after 3 , 6 12 and 24 month of the surgery
  kg of lean mass will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)

CONTACTS AND LOCATIONS:
Overall Officials: Fernández-Lao, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - Carolina Fernández Lao, Granada
  - Carolina Fernández-Lao, Granada